CLINICAL TRIAL: NCT01894126
Title: Mobile Phone One Way Short Message Service (SMS) Versus SMS Dialogue for Women's and Child Health (Mobile WACh) in Kenya: A Randomized Control Trial
Brief Title: Mobile Phone Messaging to Improve Women's and Children's Health (Mobile WACh) in Kenya
Acronym: Mobile WACh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Nairobi (Other); Kenyatta National Hospital (Other Government)
Responsible Party: Principal Investigator, Jennifer Unger, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K12HD001264-14UNGER; K12HD001264-14 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Maternal Health; Neonatal Health; Family Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Two-way SMS dialogue (Experimental): Women will receive SMS messages with prompts to reply. They will have the ability to text back to the system and both respond to and initiate SMS dialogue
  Interventions: Behavioral: Two-way SMS Dialogue
- One-way SMS Messaging (Experimental): Women will receive scheduled one-way SMS messages
  Interventions: Behavioral: One-way SMS Messaging
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Two-way SMS Dialogue
  Arms: Two-way SMS dialogue
Behavioral: One-way SMS Messaging
  Arms: One-way SMS Messaging

SUMMARY:
With the increased prevalence of cellular phones, mobile technology provides an important tool to reach underserved populations in low to middle income countries. mHealth interventions offer promise to improve maternal child health throughout the reproductive health continuum if they contribute to increasing skilled birth attendance, family planning and exclusive breastfeeding. We propose a randomized clinical trial to determine effect of using mobile phones to deliver SMS (one-way) versus an interactive SMS dialogue (two-way) on uptake of reproductive and neonatal health services and maternal and infant outcomes

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Access to a mobile phone
* Able to read SMS messages
* Willing to receive SMS messages

Exclusion Criteria:

* Unwilling or unable to meet inclusion criteria

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Contraceptive uptake | 10 weeks postpartum; 24 weeks postpartum
Facility Delivery | Postpartum
Exclusive Breastfeeding | 24 weeks postpartum

SECONDARY OUTCOMES:
ANC attendance | Postpartum
Infant Immunizations | Six months postpartum
Maternal mortality | 6 months postpartum
Infant mortality | Six months postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Mathare North Health Centre, Nairobi, Kenya

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276